CLINICAL TRIAL: NCT06909890
Title: The Effectiveness of a Natural Aqueous Extract of Chios Mastic in the Management of Dyspepsia: the MASTIQUA-D Randomized Controlled Clinical Trial
Brief Title: A Study of Chios Mastic Water in Dyspepsia
Acronym: MASTIQUA-D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Responsible Party: Principal Investigator, GIANNIS ARNAOUTIS, Assistant Professor, Harokopio University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 470/05-02-2025
Record Dates: First submitted 2025-03-21; First posted 2025-04-04 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Dyspepsia
Keywords: Pistacia Lentiscus var. Chia; Chios mastic; dyspepsia; gastrointestinal health
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): This arm will consume 600 mL of a sparkling beverage enriched with Chios mastic per day for a 3-month period.
  Interventions: Behavioral: Chios mastic beverage
- Control group (Placebo Comparator): This arm will consume 600 mL of a standard sparkling beverage per day for a 3-month period.
  Interventions: Behavioral: Placebo beverage

INTERVENTIONS:
Behavioral: Chios mastic beverage — Participants of this intervention arm will be provided with a sparkling beverage enriched with the natural mastic aqueous extract (0.2%), a by-product of Chios mastic processing, and will be asked to consume it daily (3 bottles of 200 mL each) for 3 months. Participants will also be instructed to maintain their usual lifestyle practices and medical treatment stable.
  Arms: Intervention group
Behavioral: Placebo beverage — Participants of this intervention arm will be provided with a placebo sparkling beverage (same organoleptic characteristics with experimental beverage but no active ingredients) and will be asked to consume it daily (3 bottles of 200 mL each) for 3 months. Participants will also be instructed to maintain their usual lifestyle practices and medical treatment stable.
  Arms: Control group

SUMMARY:
Chios mastic is a natural product with strong antimicrobial, anti-inflammatory and antioxidant properties, and well-established benefits for dyspeptic disorders. The aim of the present study is to investigate the effectiveness of a natural aqueous extract of Chios mastic (mastic water), a by-product of Chios mastic processing, in the management of dyspepsia. This will be a 3-month randomized double-blind controlled clinical trial in adults with dyspepsia. Participants will be blindly randomized to an intervention group, which will receive 600 mL/d of a carbonated beverage enriched with Chios mastic water (0.2%), or a control group, which will receive 600 mL/d of an identical placebo beverage with no active ingredients. Participants will be evaluated in terms of anthropometric indices, lifestyle habits, severity of dyspepsia-related gastrointestinal symptoms, quality of life, as well as biochemical markers, both pre- and post-intervention.

DETAILED DESCRIPTION:
The term "dyspepsia" encompasses a wide range of upper gastrointestinal symptoms, including early satiety, abdominal pain, flatulence, bloating, postprandial fullness or discomfort, nausea, vomiting, and heartburn. These symptoms are common in several gastrointestinal diseases and affect up to 40% of the population worldwide. Dyspepsia leads to reduced quality of life, functionality, and productivity, and has a significant detrimental impact on healthcare systems due to repeated patient visits to healthcare professionals and unnecessary prescription and use of medications.

Several natural plant products have emerged as potential therapeutic agents, due to their high content of bioactive compounds that can inhibit the manifestation of pathophysiological processes. Chios mastic is the resin of the mastic tree (Pistacia Lentiscus var. Chia), produced exclusively in the southern part of the Greek island of Chios. References about the medical use of Chios mastic from Greek populations for the treatment of gastrointestinal disorders or as a cosmetic agent can be found in ancient texts. Nowadays, this versatile resin has been rediscovered, not only as a traditional remedy and aromatic agent, but also as a potent phytotherapeutic product with strong anti-inflammatory and anti-oxidant properties. In 2015, Chios mastic was recognized as an herbal medicinal product by the European Medicines Agency (EMA), with two therapeutic indications: mild dyspeptic disorders and skin inflammation/healing of minor wounds (EMA/HMPC/46758/2015).

Over the last years, Chios mastic has been widely used in medicinal products and food supplements, and has become the object of intense study in the fields of Nutrition and Pharmacotechnology with the aim of investigating its beneficial effects on pathological conditions mainly located in the gastrointestinal system. The few available randomized controlled clinical trials in the field have mainly investigated the effect of supplemental administration of Chios mastic in patients with inflammatory bowel diseases (Crohn's disease), irritable bowel syndrome and functional dyspepsia, highlighting its benefits in reducing the severity of gastrointestinal symptoms and improving quality of life. However, no study to date has focused on the integration of a food/beverage enriched with Chios mastic into the usual diet of individuals with gastrointestinal disorders and on investigating its potential beneficial effects on gastrointestinal health, symptoms and health-related quality of life.

Given the beneficial effect of Chios mastic on gastrointestinal health, the aim of the present study is to investigate the effect of beverages, without added sugars or artificial sweeteners and enriched with natural aqueous extract of Chios mastic (mastic water), in individuals with dyspepsia. The research hypothesis is that the incorporation of beverages enriched with mastic water into the diet of individuals with dyspepsia will lead to an improvement in the severity of gastrointestinal symptoms and associated quality of life, highlighting them as functional substitutes for conventional beverages.

The study will be a 3-month parallel, randomized (allocation ratio 1:1), controlled, double-blind clinical trial in a sample of 60 adult patients with dyspepsia. Participants will be excluded on the basis of the presence of other chronic gastrointestinal diseases, the presence of other serious comorbidities, or recent significant changes in lifestyle habits. Participants will be randomized to an intervention group (IG) or a control group (CG). The IG will be provided with 600 mL of a sparkling beverage (Mastiqua lemon lime) containing the natural mastic aqueous extract (0.2%) to be consumed daily (3 bottles of 200 mL each). The CG will be provided with the same quantity of a placebo sparkling beverage, which will be identical in appearance and organoleptic characteristics, including the characteristic Chios mastic aroma. Randomization will be performed by an investigator with no clinical involvement, while all patients and study team members will be blinded to patient allocation in study groups. All enrolled patients will be asked to maintain their usual dietary and physical activity practices and keep their standard medical treatment stable throughout the study. The study physician will systematically record potential side-effects and will be in charge of terminating the intervention if needed.

At baseline and at the end of the 3-month study, participants will be evaluated in terms of anthropometric indices (body weight, height and waist circumference), body composition, lifestyle (diet and physical activity) habits, the presence and severity of dyspepsia-related gastrointestinal symptoms and quality of life. In addition, 12-h fasting blood samples will be collected and various biochemical markers (e.g., glucose metabolism indices, lipidemic profile, liver enzymes and inflammatory markers) will be measured in serum/plasma samples both pre- and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-60 years old.
* Body mass index of 20-35 kg/m2.
* Presence of dyspepsia.

Exclusion Criteria:

* Presence of chronic diseases (e.g. diabetes mellitus, cancer, cardiovascular, hepatic, renal, respiratory, chronic inflammatory and psychiatric diseases).
* Presence of other chronic gastrointestinal diseases (e.g. gastroesophageal reflux, inflammatory bowel disease and celiac disease).
* Use of immunosuppressants, anti-inflammatories, antibiotics and corticosteroids.
* Use of dietary supplements or other products with Chios mastic.
* Excessive alcohol consumption (>210 g and >140 g of ethanol per week for men and women, respectively).
* Currently on a weight-loss diet or recent (within 6 months) significant change in lifestyle habits.
* Pregnancy or breast feeding (for women)

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in dyspepsia symptoms severity | 0 (baseline) and 12 weeks
  Dyspepsia symptoms will be assessed through the Patient Assessment of Gastrointestinal Disorders - Dyspepsia Symptom Severity Index (PAGI-SYM). The questionnaire's score ranges from 0 to 100, with higher values indicating more severe symptoms.

SECONDARY OUTCOMES:
Change in quality of life | 0 (baseline) and 12 weeks
  Quality of life will be assessed through the short-form 36-item health survey (SF-36) questionnaire. SF-36 includes 2 generic scales, i.e. the Physical Component Summary and the Mental Component Summary, both ranging from 0 to 100, with 0 representing the worst possible state of health and 100 representing the optimal state of health.
Change in quality of life | 0 (baseline) and 12 weeks
  Quality of life will be assessed through the short-form 10-item Nepean Dyspepsia Index (SF-NDI) questionnaire. SF-NDI includes 5 sub-scales, i.e. tension, interference with daily activities, eating/drinking, knowledge/control and work/study, each ranging from 2 to 10, with 2 representing the highest quality of life and 10 representing the lowest quality of life.
Change in high-sensitivity C-reactive protein | 0 (baseline) and 12 weeks
  High-sensitivity C-reactive protein (mg/L) will be measured in blood samples by nephelometry.

CONTACTS AND LOCATIONS:
Overall Officials: Giannis Arnaoutis, PhD, Principal Investigator — Department of Nutrition and Dietetics, School of Health Sciences and Education, Harokopio University of Athens; Labros Sidossis, PhD, Study Director — Department of Nutrition and Dietetics, School of Health Sciences and Education, Harokopio University of Athens
Locations (1):
- Department of Nutrition and Dietetics, School of Health Sciences and Education, Harokopio University of Athens, Kallithea, Attica, Greece

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be shared to investigators for the purpose of data meta-analysis, provided that the proposed use of the data has been approved by the Study Principal Investigator. Proposals should be directed to garn@hua.gr.